CLINICAL TRIAL: NCT03400865
Title: The Effect of Combined Treatment of Cabergoline With Hydroxychloroquine/Chloroquine for Resistant Prolactinomas
Brief Title: Cabergoline Combined Hydroxychloroquine/Chloroquine to Treat Resistant Prolactinomas
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhebao Wu (Other)
Collaborators: Xinqiao Hospital of Chongqing (Other); First Hospital of China Medical University (Other); Beijing Tiantan Hospital (Other); First Affiliated Hospital of Wenzhou Medical University (Other); First Affiliated Hospital of Fujian Medical University (Other); Peking Union Medical College Hospital (Other); Huashan Hospital (Other); Chinese PLA General Hospital (Other)
Responsible Party: Sponsor-Investigator, Zhebao Wu, Chief Physician, Ruijin Hospital
Organization: Ruijin Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCCT-2018
Record Dates: First submitted 2018-01-08; First posted 2018-01-17 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-01

CONDITIONS: Resistance, Disease; Prolactinoma
Keywords: cabergoline; prolactinomas; resistant; hydroxychloroquine; chloroquine
MeSH Terms: conditions — Disease Resistance; Prolactinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HCQ/CQ and CAB combined treatment (Experimental): Subjects are treated with hydroxychloroquine sulfate tablets 5mg/kg Bid and cabergoline tablets 2mg/week for 3 months.
  Interventions: Drug: HCQ/CQ and CAB combined treatment

INTERVENTIONS:
Drug: HCQ/CQ and CAB combined treatment — Subjects are treated with hydroxychloroquine sulfate tablets 5mg/kg Bid and cabergoline tablets 2mg/week for 3 months.After therapy of 3 months the medication will be stopped if does not reduce prl level more than 20% or failure to decrease prolactinoma size.
  Other Names: HCCT

SUMMARY:
The purpose of this study is to preliminarily evaluate the safety and efficacy of cabergoline combined hydroxychloroquine/chloroquine(HCQ/CQ) therapy for cabergoline-Resistant Prolactinomas

DETAILED DESCRIPTION:
The dopamine agonist cabergoline (CAB) has been used widely in the treatment of prolactinomas, but its clinical use is hampered by intolerance and/or resistant in some patients with prolactinoma. Chloroquine (CQ) is an old drug widely used to treat malaria. Recent studies, including our own (J Clin Endocrinol Metab, 2017; Autophagy, 2017; Oncotarget, 2015), have revealed that CAB and CQ are involved in induction of autophagy and activation of autophagic cell death. Furthermore, CQ enhanced suppression of cell proliferation by CAB. We established a low-CAB-dose condition in which CAB was able to induce autophagy but failed to suppress cell growth. Addition of CQ to low-dose CAB blocked normal autophagic cycles and induced apoptosis, evidenced by the further accumulation of p62/caspase-8/LC3-II. The data suggest that combined use of CAB and CQ may increase clinical effectiveness in treatment of intolerance and/or resistant prolactinomas.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 70 years old, either sex;
2. Karnofsky performance status ≥ 70;
3. Patients who were suffered drug-resistant,which has taken cabergoline ≥2.0mg/week no less than 3 months, referring to failure to normalize PRL levels and failure to decrease macroprolactinoma size by >or=50%;
4. The patient has signed the informed consent.

Exclusion Criteria:

1. Patients concomitantly taking the psychotropic drugs or other drugs causing elevated PRL ;
2. Patients with parkinson disease and is taking dopaminergic agents;
3. Patients with prolactinoma who received Gamma knife treatment;
4. Patients who use any dopamine receptor agonists other than cabergoline;
5. pregnant or lactating women, or women preparing pregnant;
6. Patients with poor compliance, who cannot implement the program strictly.
7. History of allergic reactions attributed to compounds of similar chemical or biologic composition to HCQ.
8. Glucose-6-phosphate dehydrogenase (G6PD) deficiency, as HCQ may cause hemolytic anemia in patients with G6PD deficiency.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-10-25 (Estimated); Primary Completion 2020-12-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline on prolactin(PRL) level | Up to 6 months
  Record the result of prolactin on every 3 month follow-up visit

SECONDARY OUTCOMES:
Change from baseline on tumor volume measured by enhanced pituitary Magnetic Resonance Imaging（MRI） | Up to 6 months
  Record the tumor volume from enhanced pituitary MRI on every 3 month follow-up visits
Change from baseline of visual acuity | Up to 6 months
  Record the Visual acuity on every 3 month follow-up visit
Change from baseline on 5 point visual field scale | Up to 6 months
  Record the Visual field scale on every 3 month follow-up visit, 0 = normal, no vision loss; 1 = one quadrant vision loss; 2 = two quadrants of vision loss; 3 = three quadrants of vision loss; 4 = four quadrants of vision loss but retain a central tubular vision; 5 = blind

CONTACTS AND LOCATIONS:
Overall Officials: Zhebao Wu, Medical, Study Chair — Ruijin Hospital
Locations (9):
- China (9):
  - Beijing Tiantan Hospital, Beijing, Beijing Municipality
  - Huashan Hospital, Shanghai, Shanghai Municipality
  - Ruijin Hosipital, Shanghai, Shanghai Municipality
  - Chinese PLA General Hospital, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Xinqiao Hospital of Chongqing, Chongqing
  - First Affiliated Hospital of Fujian Medical, Fujian
  - First Hospital of China Medical University, Shenyang
  - First Affiliated Hospital of Wenzhou Medical Univeristy, Wenzhou

IPD SHARING:
Plan to Share IPD: Undecided
The individual patient Data would not be shared to the third facility, but the sponsor hasn't decided whether to share the individual patient date to the other related studies hold by himself in the future.

REFERENCES:
- [Background] Leng ZG, Lin SJ, Wu ZR, Guo YH, Cai L, Shang HB, Tang H, Xue YJ, Lou MQ, Zhao W, Le WD, Zhao WG, Zhang X, Wu ZB. Activation of DRD5 (dopamine receptor D5) inhibits tumor growth by autophagic cell death. Autophagy. 2017 Aug 3;13(8):1404-1419. doi: 10.1080/15548627.2017.1328347. Epub 2017 Jun 14. PMID 28613975
- [Background] Lin SJ, Leng ZG, Guo YH, Cai L, Cai Y, Li N, Shang HB, Le WD, Zhao WG, Wu ZB. Suppression of mTOR pathway and induction of autophagy-dependent cell death by cabergoline. Oncotarget. 2015 Nov 17;6(36):39329-41. doi: 10.18632/oncotarget.5744. PMID 26513171
- [Result] Lin SJ, Wu ZR, Cao L, Zhang Y, Leng ZG, Guo YH, Shang HB, Zhao WG, Zhang X, Wu ZB. Pituitary Tumor Suppression by Combination of Cabergoline and Chloroquine. J Clin Endocrinol Metab. 2017 Oct 1;102(10):3692-3703. doi: 10.1210/jc.2017-00627. PMID 28973192